CLINICAL TRIAL: NCT03290573
Title: Site Selection of Peripheral Venous Access Via Short Peripheral Catheters in Adult Patients (SPECIAL Trial)
Brief Title: Site Selection of Short Peripheral Venous Catheters
Acronym: SPECIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Chuanjie Wu, MD, PhD, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FAHZU-2017-016
Record Dates: First submitted 2017-09-17; First posted 2017-09-25 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Short Peripheral Venous Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dorsum of hand group (Active Comparator): short peripheral venous catheter place in the dorsum of the hand
  Interventions: Device: short peripheral venous catheter
- Forearm group (Experimental): short peripheral venous catheter place in the forearm
  Interventions: Device: short peripheral venous catheter

INTERVENTIONS:
Device: short peripheral venous catheter — short peripheral venous catheter for infusion therapy in adult patients

SUMMARY:
Up to 90% of catheters fail before therapy is complete. Improved dwell time of intravenous catheters for even small increments of time would further reduce the number of insertions, staff workloads, and costs. In this study, the investigators investigated whether short peripheral venous catheter site of insertion influence the dwell time.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Expected duration of infusion therapy by short peripheral intravenous catheters >7 days
* Give written informed consent

Exclusion Criteria:

* The peripheral venous catheter was inserted in emergency room or in emergency circumstances
* Bloodstream infection
* Had a peripheral venous catheter already in situ at the baseline
* Altered mental state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1517 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2019-01-06 (Actual)

PRIMARY OUTCOMES:
Indwelling time | from the cannulae insertion until its removal, usually within 2 weeks

SECONDARY OUTCOMES:
Phlebitis | from the cannulae insertion until its removal, usually within 2 weeks
Occlusion of the catheter | from the cannulae insertion until its removal, usually within 2 weeks
Infiltration | from the cannulae insertion until its removal, usually within 2 weeks
Accidental catheter removal | from the cannulae insertion until its removal, usually within 2 weeks
Local venous infection | from the cannulae insertion until its removal, usually within 2 weeks
Catheter-related bloodstream infection | from the cannulae insertion until its removal, usually within 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjie Wu, MD, Study Chair — The First Affiliated Hospital of Zhengzhou University
Locations (6):
- China (6):
  - Suzhou municipal hospital, Suzhou, Anhui
  - Xuanwu Hospital Captial Medical University, Beijing, Beijing Municipality
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangtan Central Hospital, Xiangtan, Hunan